CLINICAL TRIAL: NCT01395979
Title: HIV Prevention and Trauma Treatment for Men Who Have Sex With Men With Childhood Sexual Abuse Histories
Acronym: THRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Fenway Community Health (Other); University of Miami (Other)
Responsible Party: Principal Investigator, Conall O'Cleirigh, Ph.D., Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH095624-01 (NIH)
Record Dates: First submitted 2011-07-11; First posted 2011-07-18 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Sexual Risk Behavior; Childhood Sexual Abuse; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Processing Therapy for Sexual Risk (CPT-SR) (Experimental): The CPT-SR condition will be comprised of 10 individual therapy sessions fully integrating sexual risk reduction counseling into cognitive therapy for sexual abuse-related trauma.
  Interventions: Behavioral: Cognitive Processing Therapy for Sexual Risk; Behavioral: Sexual Risk Reduction Intervention
- Time-Matched Control (TMC) (Active Comparator): The TMC will be comprised of sexual risk reduction counseling/education and supportive psychotherapy.
  Interventions: Behavioral: Supportive Psychotherapy; Behavioral: Sexual Risk Reduction Intervention

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy for Sexual Risk — Eight weekly sessions, 4 modules.
  Other Names: CPT-SR
  Arms: Cognitive Processing Therapy for Sexual Risk (CPT-SR)
Behavioral: Supportive Psychotherapy — Eight weekly sessions
  Other Names: TMC
  Arms: Time-Matched Control (TMC)
Behavioral: Sexual Risk Reduction Intervention — Two weekly sessions.

SUMMARY:
Brief Summary: The specific aims of this study are:

1. To test, in a two-arm randomized controlled trial, the efficacy of cognitive processing therapy for sexual risk and posttraumatic symptom severity reduction (CPT-SR) in HIV-uninfected men who have sex with men (MSM) who have histories of childhood sexual abuse (CSA). The primary outcome is reduction in unprotected anal/vaginal intercourse (number and proportion) with serodiscordant partners. The investigators will also examine the intervention effect on CSA-related trauma symptom severity and cognitions and behaviors.
2. To examine the degree to which intervention-related reductions in sexual risk behavior are mediated by reductions in CSA-related symptom severity, cognitions, and behaviors.
3. To examine the degree to which the intervention reduces incident sexually transmitted infections (STIs) during the study period, as well as to explore additional potential moderators and mediators of intervention efficacy.

Study hypotheses:

1. For the primary outcome, the investigators hypothesize that those who receive the intervention will have reduced transmission-risk behavior.
2. For the secondary outcome, the investigators hypothesize that those who receive the intervention will have reduced trauma symptom severity (cognitions and behaviors).

DETAILED DESCRIPTION:
The prevalence of HIV among men who have sex with men (MSM) is estimated at an alarming 19% domestically (CDC 2010), rates comparable to endemic settings in certain regions of sub-Saharan Africa where approximately 20% of the adult population is HIV infected. Studies have also demonstrated a staggeringly high prevalence of childhood sexual abuse (CSA) in MSM, and shown an association between CSA and HIV risk in MSM. A successful intervention for MSM with a CSA history to prevent HIV has the potential to avert infections among some of the riskiest members of the most HIV vulnerable group in the U.S. Notwithstanding the ability of the existing HIV prevention interventions to show reductions in sexual risk taking, the recent successes of chemoprophylaxis, current policy initiatives, and empirically supported recommendations, all support development of combination prevention interventions that can specify multiple prevention targets, address related risk factors and barriers, and are grounded in a community context. The pathways from CSA to adult sexual risk behavior are varied and complex and this complexity is appropriately addressed in individual-based interventions where empirically supported interventions for CSA related trauma were efficacy tested. The development of an integrated prevention intervention that utilizes cognitive behavioral technologies to address co-occurring and interfering CSA and sexual risk represents a novel and largely untested innovative application that is theoretically designed to address sexual risk directly and indirectly through reductions in CSA-related trauma symptoms. The flexibility of integrated and combination prevention programs has the potential to support triage of MSM with particular risk profiles to the programs that best meet their prevention needs.

This two-arm RCT is designed to test the efficacy of a psycho-social intervention that addresses intersecting epidemics among MSM, HIV and CSA. The experimental condition integrates sexual risk reduction counseling with Cognitive Processing Therapy for Sexual Risk (CPT-SR). CPT-SR has been specifically piloted on MSM with CSA histories and sexual risk to reduce interfering negative CSA-related thoughts about self, to more accurately appraise sexual risk, and to decrease avoidance of sexual safety considerations through rehearsals of sexual safety behaviors. The active and time-matched comparison condition is risk reduction counseling plus supportive psychotherapy. The investigators will randomize HIV-uninfected MSM who report a history of CSA and multiple recent sexual risk episodes for HIV (unprotected anal/vaginal intercourse) across two sites (Boston and Miami). The primary outcome will be self-reported sexual risk taking as assessed via a computer-based questionnaire. Secondary outcomes include trauma symptom severity, both cognitive and behavioral. Study assessment points are at baseline, 3 (post treatment), 6, 9, and 12-month follow-ups.

ELIGIBILITY:
Eligibility Criteria:

Inclusion Criteria:

* Identifies as MSM.
* Reports history of CSA (sexual contact before the age of 13 with an adult or person 5 years older or sexual contact with the threat of force or harm between the ages of 13 and 16 inclusive or with a person 10 years older).
* Reports >1 episode of unprotected anal or vaginal intercourse within the past three months.
* Reports HIV-negative status confirmed by rapid HIV test.
* Is capable of completing and fully understanding the informed consent process and the study procedures.

Exclusion Criteria:

* All episodes of unprotected anal or vaginal intercourse occurred with only a single, primary HIV-negative partner.
* Significant mental health diagnosis requiring immediate treatment (e.g. bipolar disorder; any psychotic disorder).
* Inability to complete informed consent process (e.g. substantial cognitive impairment, inadequate English language skills).
* Has received CPT for PTSD within the past 12 months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in Sexual Risk Behavior for HIV Acquisition | Baseline, (2 weeks post-baseline pre-randomization), 3,6, 9, and 12 month follow ups
  Number of unprotected (no condom was used) insertive or receptive anal or vaginal intercourse acts reported in the past 3 months with casual partners or with partners with unknown or positive HIV status.

SECONDARY OUTCOMES:
Changes from Baseline in Trauma Symptom Severity | Baseline assessment, 3, 6, and 9-month follow-up assessments
  Davidson Trauma Scale which has been correlated with measures of Post-Traumatic Stress Disorder (PTSD) severity, depression, and general anxiety, and discriminated well between traumatized individuals with and without PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: Conall O'Cleirigh, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - University of Miami, Coral Gables, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Fenway Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Batchelder AW, Fitch C, Feinstein BA, Thiim A, O'Cleirigh C. Psychiatric, Substance Use, and Structural Disparities Between Gay and Bisexual Men with Histories of Childhood Sexual Abuse and Recent Sexual Risk Behavior. Arch Sex Behav. 2021 Oct;50(7):2861-2873. doi: 10.1007/s10508-021-02037-1. Epub 2021 Oct 21. PMID 34676467
- [Derived] Batchelder AW, Choi K, Dale SK, Pierre-Louis C, Sweek EW, Ironson G, Safren SA, O'Cleirigh C. Effects of syndemic psychiatric diagnoses on health indicators in men who have sex with men. Health Psychol. 2019 Jun;38(6):509-517. doi: 10.1037/hea0000724. Epub 2019 Apr 11. PMID 30973745